CLINICAL TRIAL: NCT05938985
Title: Psychometric Properties of the Croatian Version of the Ocular Surface Disease Index Questionnaire
Brief Title: Croatian Version of the Ocular Surface Disease Index Questionnaire (OSDI)
Acronym: Cro-OSDI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Karla Randelovic, Study Coordinator, Ophthalmology Consultant, University Hospital Sestre Milosrdnice
Other Study IDs: 251-29-11-23-03
Record Dates: First submitted 2023-06-10; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with dry eye disease (DED): DED diagnosis defined by the Dry Eye Workshop (DEWS) II.
  Interventions: Diagnostic Test: Questionnaires and dry eye tests
- control (non-DED): No significant ocular disease other than refractive error and no systemic disease likely to be associated with dry eye. The non-DED group will be sex-matched and age-matched to the DED patients.
  Interventions: Diagnostic Test: Questionnaires and dry eye tests

INTERVENTIONS:
Diagnostic Test: Questionnaires and dry eye tests — Ocular Surface Disease Index (OSDI), National Eye Institute Visual Functioning Questionnaire (NEI VFQ-25), best visual acuity (BCVA) measuring, intraocular pressure, corneal fluorescein staining, lissamine green staining, Schirmer test type I and II, tear breakup time (TBUT) and noninvasive tear breakup time (NIBUT).

SUMMARY:
Ocular Surface Disease Index (OSDI) Questionnaire is an important tool for the diagnosis of dry eye disease. Croatian version is yet not available. With a permission of AbbVie company investigators want to make a Croatian version of the Ocular Surface Disease Index Questionnaire (Cro-OSDI).

DETAILED DESCRIPTION:
Aim is to translate, adapt and validate the Croatian version of the Ocular Surface Disease Index (OSDI) Questionnaire. Validation process of the Croatian version of the OSDI questionnaire will be accomplished in two phases: the translation and assessment of psychometric properties.

The translation process will involve the following steps based on the previously established guidelines. First is forward translation, the second is backward translation and the third is pilot study. The final version (the Cro-OSDI) will be used to test psychometric properties of the Croatian version of the questionnaire.

Eligible participants will complete the Cro-OSDI and and the previously validated Croatian version of the National Eye Institute Visual Functioning Questionnaire (NEI VFQ-25). After completing the respective questionnaires, the participants will undergo a complete ophthalmic examination for both eyes and dry eye tests (corneal fluorescein staining, lissamine green staining, Schirmer test type I and II, tear break-up time (TBUT), noninvasive tear breakup time (NIBUT)).

ELIGIBILITY:
Inclusion Criteria:

* native Croatian-speaking participants with normal cognitive ability
* DED diagnosis complied with those defined by the DEWS II
* DED for at least 3 months
* BCVA logMAR< 0.6 or better

Exclusion Criteria:

* symptoms of conjunctivitis
* a history of contact lens use
* previous intraocular or ocular surface surgeries within the previous 6 months
* allergies
* eyelid malpositions
* ptosis
* Parkinson disease
* hereditary corneal disease
* any other disease that could affect blinking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that are coming for an examination to an ophthalmology department of University Hospital.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-02 (Estimated)

PRIMARY OUTCOMES:
OSDI translation to the Croatian language and Cro-OSDI score measurement | 2 weeks
  Ocular Surface Disease Index will be first translated into Croatian language in forward and backward manner. Further on, translated (Cro-OSDI) will be conducted on population of selected participants, and the Cro-OSDI score will be determined. OSDI score is in a range from normal (0-12 points) till severe dry eye (33-100 points).

SECONDARY OUTCOMES:
Cro-OSDI score comparison with the NEI VFQ-25 score | 2 months
  Cro-OSDI score that was measured as a Primary measure will then be compared with the translated and standardized score NEI VFQ-25 score, which will serve as a validation test for the translated Cro-OSDI score. In National Eye Institute Visual Functioning Questionnaire, 100 is the best score and 0 is the worst score.
Cro-OSDI score comparison with the Oxford scale, SICCA scale, scaled filter paper strips. | 2 months
  Cro-OSDI score that was measured as a Primary measure will then be compared with the dry eye clinical tests (corneal fluorescein staining scale from absent (0) to severe(5), lissamine green staining scale from 0-3 scale based on scale density, Schirmer test type I (under 5 mm is dry eye) and II (under 10 mm is dry eye), tear breakup time (TBUT, under 7 seconds is dry eye) and noninvasive tear breakup time (NIBUT-under 8 seconds is dry eye). This will serve as a validation procedure for the translated Cro-OSDI score.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided